CLINICAL TRIAL: NCT03845881
Title: A Randomized, Double-Blinded, Placebo-Controlled Trial Comparing a Multi-Modal Pain Protocol With and Without Opioids Following Total Joint Arthroplasty
Brief Title: Trial Comparing a Multi-Modal Pain Protocol With and Without Opioids Following Total Joint Arthroplasty
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Ambit Biosciences Corporation (Industry); Kern Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin K. Wilke, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 18-004256
Record Dates: First submitted 2019-02-11; First posted 2019-02-19 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Intervention Model Description: Multi-Modal Pain Protocol with and without Opioids Following Total Joint Arthroplasty
Who Masked: Participant, Investigator
Masking Description: The oxycodone and placebo tablets will be encapsulated by the research pharmacy prior to dispensing for blinding purposes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid (Active Comparator): Multi-Modal Pain Protocol with Opioids Following Total Joint Arthroplasty
  Interventions: Drug: Oxycodone
- Non Opioid (Placebo Comparator): Multi-Modal Pain Protocol without Opioids Following Total Joint Arthroplasty
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Oxycodone — The primary endpoint will be pain scores, calculated by the Visual Analog Scale. This score will be collected daily during the hospital examination and by phone surveys for two weeks following discharge. Investigators hypothesize that the non-opioid pain regimen will provide equivalent relief as compared to the opioid regimen.
  Arms: Opioid
Drug: Placebo Oral Tablet — The primary endpoint will be pain scores, calculated by the Visual Analog Scale. This score will be collected daily during the hospital examination and by phone surveys for two weeks following discharge. Investigators hypothesize that the non-opioid pain regimen will provide equivalent relief as compared to the opioid regimen.
  Arms: Non Opioid

SUMMARY:
To help curb the use of opioid medications following orthopedic surgery investigators have developed a new multi-modal pain pathway. Investigators aim to compare this regimen with and without the inclusion of opioid medications. This study will be performed in a randomized, double-blinded, placebo-controlled fashion in patients undergoing primary total knee or total hip arthroplasty. Investigators hypothesize that the opioid devoid pathway will show equivalent pain scores to the pathway that includes opioids while also having less constipation, nausea, and vomiting following surgery. If successful, this would create a dramatic decrease in opioid consumption following orthopedic surgery while still providing appropriate pain relief to patients.

DETAILED DESCRIPTION:
* Aim 1 will be to compare the postoperative pain levels both in the hospital setting as well as daily for two weeks following discharge between patients in the opioid treatment group and those in the non-opioid treatment group. This will be performed with clinical exams while in the hospital and with phone surveys on discharge. Results will be recorded using the Visual Analog Scale for pain scores.
* Aim 2 will be to compare the overall morphine equivalents used during hospitalization between the opioid and non-opioid treatment groups. This will be calculated based on the amount of intravenous breakthrough narcotic pain medication used in the hospital setting (divided by the total number of post-surgery hospitalization hours to account for varying lengths of stay). Investigators will also measure the total number of opioid pills (these would be placebo pills for the non-opioid group) consumed during the first two weeks post-discharge, and the post-surgery day on which opioid pills were discontinued, and compare these outcomes between the opioid and non-opioid groups.
* Aim 3 will be to compare postoperative constipation, nausea, and vomiting between the two treatment groups. This will be assessed with daily clinical examinations while in the hospital and with daily phone surveys on discharge. Constipation will be recorded as presence or absence, while nausea and vomiting will be measured using the Postoperative Nausea and Vomiting Scale.
* Aim 4 will be to compare the length of post-surgery hospitalization between the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 and < 90 years.
2. Willing to participate in the study and competent to provide informed consent.
3. Willing to comply with protocol procedures.
4. Has an underlying diagnosis of osteoarthritis indicated for knee arthroplasty.

Exclusion Criteria:

1. A diagnosis of renal or liver disease
2. If a patient has a contraindication to receiving a spinal anesthetic or pain catheter
3. The patient must not have taken any narcotic medications during the 3 months leading up to the surgery
4. The patient must not be allergic or intolerant to a medication used in the multi-modal pain pathway
5. Revision hip or knee arthroplasty
6. If a patient is being treated under worker's compensation
7. If a patient has diabetes
8. Unable to take Aspirin 325 mg twice daily for deep venous thromboprophylaxis

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
Pain Levels | 2 weeks
  compare the postoperative pain levels both in the hospital setting as well as daily for two weeks following discharge between patients in the opioid treatment group and those in the non-opioid treatment group. This will be performed with clinical exams while in the hospital and with phone surveys on discharge. Results will be recorded using the Visual Analog Scale for pain scores. This scale ranges from 0 to 10, with zero being no pain and 10 being as bad as can be, and includes visual facial cues. Following this scale, investigators will also ask about sleep, activity, mood, and stress.

SECONDARY OUTCOMES:
Opioid Levels | 2 weeks
  compare the overall morphine equivalents used during hospitalization between the opioid and non-opioid treatment groups. This will be calculated based on the amount of intravenous breakthrough narcotic pain medication used in the hospital setting (divided by the total number of post-surgery hospitalization hours to account for varying lengths of stay). Investigators will also measure the total number of opioid pills (these would be placebo pills for the non-opioid group) consumed during the first two weeks post-discharge, and the post-surgery day on which opioid pills were discontinued, and compare these outcomes between the opioid and non-opioid groups.
Side effects | 2 weeks
  compare postoperative constipation, nausea, and vomiting between the two treatment groups. This will be assessed with daily clinical examinations while in the hospital and with daily phone surveys on discharge. Constipation will be recorded as presence or absence, while nausea and vomiting will be measured using the Postoperative Nausea and Vomiting Scale. This scaled is based off 2 questions related to nausea and vomiting which will be added together for a total score. Responses range from 0 to 3 and a total score of greater than or equal to 5 will be defined as clinically important.
Length of hospitalization | 2 weeks
  compare the length of post-surgery hospitalization between the two treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Wilke, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials